CLINICAL TRIAL: NCT01748045
Title: The Use of Inhaled Nitric Oxide to Improve Respiratory Outcomes in Late Preterm Infants
Brief Title: Study of Inhaled Nitric Oxide (iNO) and Respiratory Outcomes in Late Preterm Infants
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Enrollenment has been suspended due to poor enrollment
Sponsor: Tufts Medical Center (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10487
Record Dates: First submitted 2012-11-20; First posted 2012-12-12 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Inhaled Nitric Oxide; Bronchopulmonary Dysplasia; Late Prematurity; Chronic Respiratory Morbidity
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Inosine; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inhaled Nitric Oxide (Experimental): iNO to start at 20 parts per million (ppm) for the first three days of life. The dose will then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Interventions: Drug: inhaled nitric oxide
- Nitrogen Gas (Placebo Comparator): Placebo gas will be adjusted the same as study gas: to start at 20ppm for the first three days of life. The dose will then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Interventions: Drug: Placebo Comparator - nitrogen gas

INTERVENTIONS:
Drug: inhaled nitric oxide
  Other Names: iNO, INOmax
  Arms: inhaled Nitric Oxide
Drug: Placebo Comparator - nitrogen gas
  Arms: Nitrogen Gas

SUMMARY:
The aim of this study is to determine if inhaled nitric oxide will improve short and long term respiratory outcomes in preterm infants. Infants born at a gestational age of 30-36 weeks and who require breathing support with high flow nasal cannula, nasal continuous positive airway pressure, or nasal intermittent positive pressure will be randomized to receive either inhaled nitric oxide or placebo. The dose will then be decreased per protocol until all respiratory support has been discontinued. Infants will be followed to evaluate safety and efficacy of non-invasive iNO delivery, up to 12 months corrected gestational age.

ELIGIBILITY:
Inclusion Criteria:

* <48 hours of age,
* 30 - 36 weeks gestational age at birth based on best estimate using obstetrical sonography (first or second trimester), solid dating criteria, or Ballard examination,
* Birth weight of ≥ 1,000 g,
* 5 minute Apgar score ≥5,
* Requiring nasal cannula O2 > 1 liter per minute (LPM), continuous positive pressure (CPAP), or non invasive positive pressure ventilation (NIPPV) for treatment of respiratory failure,
* Requiring a fraction of inspired oxygen (FIO2) of at least 0.25 to maintain arterial oxygen saturation (SaO2) 88-94%,
* Parent or guardian has signed informed consent and agrees to all study- related procedures, including those required after hospital discharge.

Exclusion Criteria:

* Major congenital anomaly
* Intubation and surfactant in the delivery room or prior to enrollment in the Neonatal Intensive Care Unit (NICU). Excludes intubation for suctioning.
* Known congenital infection (bacterial, viral),
* Perinatal asphyxia (5 minute Apgar <5, umbilical artery pH < 7.0 or evidence of neonatal encephalopathy),
* Mother and/or infant is enrolled in another clinical trial (excluding observational) or has received an investigational drug,
* Has undergone or is anticipated to require a major surgical procedure within the first 48 h of life,
* Any condition which could preclude receiving study drug or performing any study-related procedures,
* Use of postnatal corticosteroids,
* Parent or guardian is unable or unwilling to complete study procedures after hospital discharge.

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W Lee, MD, MS, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled Nitric Oxide (iNO): Number of participants who have started on iNO at 20 parts per million (ppm) for the first three days of life. The dose was then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  inhaled nitric oxide
- Nitrogen Gas: Number of participants who have started on placebo gas that was adjusted the same as study gas: to start at 20ppm for the first three days of life. The dose was decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Placebo Comparator - nitrogen gas
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide (iNO) | Nitrogen Gas
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inhaled Nitric Oxide: iNO to start at 20ppm for the first three days of life. The dose will then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  inhaled nitric oxide
- Nitrogen Gas: Placebo gas will be adjusted the same as study gas: to start at 20ppm for the first three days of life. The dose will then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Placebo Comparator - nitrogen gas
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: days] | 1 (0) | 1 (0) | 1 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Alive Without the Need for Intubation or Mechanical Ventilation Within the First Week of Life
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Inhaled Nitric Oxide: Number of participants who were started on inhaled Nitric Oxide (iNO) at 20 parts per million (ppm) for the first three days of life. The dose was then decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  inhaled nitric oxide
- Nitrogen Gas: Number of participants who were started on placebo gas that was adjusted the same as study gas: to start at 20ppm for the first three days of life. The dose was then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Placebo Comparator - nitrogen gas
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

2. Secondary Outcome: Number of Participants Who Had the Need for Exogenous Surfactant
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Inhaled Nitric Oxide: Number of participants who have started on iNO at 20ppm for the first three days of life. The dose was then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  inhaled nitric oxide
- Nitrogen Gas: Number of participants who have started on placebo gas that was adjusted the same as study gas: to start at 20ppm for the first three days of life. The dose was then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Placebo Comparator - nitrogen gas
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

3. Secondary Outcome: Total Length of Hospital Stay
Description: participants who were followed for the duration of hospital stay
Time Frame: From hospital admission through discharge
Measure: Mean (Standard Deviation); unit: days
Groups:
- Nitrogen Gas: Number of participants who have started on placebo gas which was adjusted the same as study gas: to start at 20ppm for the first three days of life. The dose was then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Placebo Comparator - nitrogen gas
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 2 | 1
days | 17.5 (2.5) | 11 (0)

4. Secondary Outcome: Total Duration of Supplemental Oxygen
Description: Participants were followed for the duration of hospital stay for use of supplemental oxygen
Time Frame: From Hospital Admission through discharge
Measure: Mean (Standard Deviation); unit: days
Groups:
- Inhaled Nitric Oxide: Number of participants who have started on iNO at 20ppm for the first three days of life. The dose were then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  inhaled nitric oxide
- Nitrogen Gas: Number of participants who have started on placebo gas will be adjusted the same as study gas: to start at 20ppm for the first three days of life. The dose were then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Placebo Comparator - nitrogen gas
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 2 | 1
days | 5 (1) | 3 (0)

5. Secondary Outcome: Diagnosis of Bronchopulmonary Dysplasia (BPD)
Description: Diagnosis of BPD by oxygen challenge test at 36 weeks post menstrual age (PMA) for infants born between 30 and 32 weeks gestational age (GA). For those born 32 1/7 - 36 weeks, an oxygen challenge test was performed at 1-2 months of age.
Time Frame: At 36 weeks postmenstrual age or 1-2month of age
Measure: Count of Participants; unit: Participants
Groups:
- Nitrogen Gas: Number of participants who have started on placebo gas was adjusted the same as study gas: to start at 20ppm for the first three days of life. The dose was then be decreased to 10 ppm for three days, 5 ppm for 3 days and then 2 ppm until all high flow respiratory support has been discontinued.
  Placebo Comparator - nitrogen gas
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

6. Secondary Outcome: Evidence of Chronic Respiratory Morbidity at 12 Months Corrected Gestational Age (CGA)
Description: defined by a validated system of parental diaries and pulmonary questionnaires, as well as review of medical records (medical visits, respiratory medication use, emergency room visits, and hospital re-admissions)
Time Frame: 12 months corrected gestational age
Population: Analysis not performed at one year corrected age, since study closed.
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

7. Secondary Outcome: Total Duration of Respiratory Support
Description: participants were followed for the duration of hospital stay for respiratory support
Time Frame: From hospital admission through discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 2 | 1
days | 5.5 (1.5) | 4 (0)

ADVERSE EVENTS:
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=2) | Nitrogen Gas (N=1)
Murmur (Cardiac disorders) | 1 (1) | 0 (0) — Infant developed a murmur consistent with peripheral pulmonic stenosis and anemia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No